CLINICAL TRIAL: NCT00798681
Title: EPICOS- Evaluating the Influence of RTU Parenteral Nutrition in the Clinical Outcome Patients Study
Brief Title: Evaluating the Influence of Ready-to-use (RTU) Parenteral Nutrition in the Clinical Outcome of Patients Study
Acronym: EPICOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fernandes Tavora Hospital (Other)
Collaborators: Hospital Bandeirantes (Other); Hospital Santa Luzia (Unknown); Hospital Samaritano (Unknown); Hospital da Polícia Militar (Unknown); Sanatório Los Arcos (Unknown); Sanatório Trinidad Palermo (Unknown); Hospital Roosevelt (Unknown)
Responsible Party: Alessandro Pontes-Arruda, MD MSc PhD FCCM, Fernandes Tavora Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HFT-001/2008-BR
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-07

CONDITIONS: Parenteral Nutrition
Keywords: parenteral nutrition; ready-to-use; customized nutrition formulation; olive oil; soybean oil; LCT/MCT; Clinoleic; oliclinomel; number of infections associated with TPN delivery system; BSI; Infection rates
MeSH Terms: conditions — Hyperphagia | interventions — Olive Oil; ClinOleic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Patients will receive RTU TPN with olive-oil as the primary source of lipids
  Interventions: Dietary Supplement: RTU TPN with olive oil as the primary lipid source
- 2 (Active Comparator): CNF parenteral nutrition made with olive oil as the primary source of lipids
  Interventions: Other: CNF Parenteral nutrition
- 3 (Active Comparator): CNF parenteral nutrition made with LCT/MCT as the primary source of lipids
  Interventions: Other: CNF parenteral nutrition

INTERVENTIONS:
Dietary Supplement: RTU TPN with olive oil as the primary lipid source — RTU will be provided as a 3 in 1 TPN ready-to-use TPN system in industrialized bags with 2.000 ml. The number of calories will be adjusted in accordance with patients' individual needs.
  Other Names: OliClinomel, Baxter Healthcare
  Arms: 1
Other: CNF Parenteral nutrition — CNF parenteral nutrition made with olive oil as the primary source of lipids
  Other Names: ClinOleic, Baxter Healthcare
  Arms: 2
Other: CNF parenteral nutrition — 3 in 1 CNF parenteral nutrition made with LCT/MCT as the primary source of lipids
  Other Names: LCT/MCT providers may vary
  Arms: 3

SUMMARY:
This is an international prospective randomized multicenter open-label controlled study. The primary center will be Fernandes Távora Hospital (Fortaleza, Ceará). The aim of this study is to investigate the effects of closed parenteral nutrition systems when compared to open parenteral nutrition systems in terms of several clinical outcomes.

DETAILED DESCRIPTION:
In most Latin-American countries individually customized nutrition formulations (CNF) remains the gold-standard for parenteral nutrition in opposition to industrialized ready-to-use parenteral nutrition (RTU). Although CNF is possibly associated with elevated infection rates, delay in the start of enteral nutrition and worse clinical outcomes there is no strong scientific evidence in the literature to support that the use of RTU is indeed associated with better clinical outcomes.

The use of closed ready-to-use parenteral nutrition systems is probably associated with less infection rates and better clinical outcomes including less time at the hospital and at the intensive care unit, less consumption of hospital resources and most likely lower mortality rates as well as early initiation of parenteral nutrition support. The aim of this study is to evaluate all the above mentioned parameters in contrast with those observed when using CNF parenteral nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with recommendation to use total parenteral nutrition.
* Caloric goals will be calculated using BEE adjusted by the pathology of the patient. In addition, patients MUST achieve at least once 75% of BEE (calculated using the Harris-Benedict equation) to be considered evaluable. Caloric intake will be accessed in a daily basis.
* This study will be performed in accordance with all ethics statements of the Helsinki's Declaration (52nd General Assembly of the World Medical Association, Edinburgh, Scotland, October, 2000), and of the Nuremberg Code.
* In addition, this study must be approved by the Institutional Review Board before patient enrollment and by the Federal Council of Research and Ethics of the Ministry of Health.
* All participating institutions will also be requested to observe Good Clinical Practice Guidelines and all federal laws and regulations.
* An informed consent will be obtained from all patients or their legal representatives before any study related procedure.

Exclusion Criteria:

* Pregnancy or breastfeeding
* Patients under 18 years of age
* Significant limitation of survival prognosis (patients expecting a life survival under 28 days due to a chronic and/or incurable disease such as uncontrolled cancer or other terminal disease)
* Pre-existing chronic renal insufficiency and need of hemodialysis or peritoneal dialysis, participation in other clinical trial less than 3 months before inclusion in this trial
* Head trauma with a Glasgow Come Score (GCS) less or equal to 5
* Severe immunologic suppression (defined as a leukocyte count bellow 5.000 cells/mm3)
* Infection by the human immunodeficiency virus
* Patients with no indication for parenteral feeding or in the imminence of receiving enteral nutrition
* Patients receiving partial parenteral nutrition in order to achieve caloric goal, or patient's, patient's legal representative or physicians decision to exclude patients from this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2008-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Incidence of bloodstreams and catheter infection, as well as incidence of sepsis, severe sepsis and septic shock. Sepsis diagnostic criteria will be re-evaluated on a daily basis. | 28-day follow up

SECONDARY OUTCOMES:
28-days all cause mortality | 28-days follow-up period
Time to start parenteral nutrition, defined as the time from prescription to the effective start of infusion | Time from prescription to the effective start of TPN
Incidence of hyperglycemic events, defined as the number of times patients developed blood glucose levels over 110 mg/dL and over 150 mg/dL | For the duration of TPN
Incidence of hypoglycemic events: defined as the number of times patients developed blood glucose levels bellow 60 mg/dL | For the duration of TPN
Mean dose of insulin used (patients will receive insulin in order to maintain blood glucose levels <150 mg/dL (or 8.3 mmol/L) in accordance with the Surviving Sepsis Campaign Guidelines) | For the duration of TPN
Use of hospital/ICU resources such as vasopressors, mechanical ventilation, need of hemodialysis, need of inotropic agents, antibiotics and sedatives | 28-days follow-up period
ICU-free days, defined as the number of days from study entry (baseline) to the actual day that a patient remained on the ICU during the 28-days follow up period | 28-days follow-up period
Number of new organ failures | 28-days follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Pontes-Arruda, MD, MSc, PhD, FCCM, Principal Investigator — Fernandes Tavora Hospital
Locations (8):
- Argentina (2):
  - Sanatorio Los Arcos, Buenos Aires
  - Sanatorio Trinidad Palermo, Buenos Aires
- Brazil (5):
  - Fernandes Tavora Hospital, Fortaleza, Ceará
  - Hospital Santa Luzia, Brasília, Federal District
  - Hospital da Polícia Militar, Rio de Janeiro, Rio de Janeiro
  - Hospital Samaritano, Rio de Janeiro, Rio de Janeiro
  - Hospital Bandeirantes, São Paulo, São Paulo
- Hospital Roosevelt, Guatemala City, Guatemala

REFERENCES:
- [Derived] Pontes-Arruda A, Dos Santos MC, Martins LF, Gonzalez ER, Kliger RG, Maia M, Magnan GB; EPICOS Study Group. Influence of parenteral nutrition delivery system on the development of bloodstream infections in critically ill patients: an international, multicenter, prospective, open-label, controlled study--EPICOS study. JPEN J Parenter Enteral Nutr. 2012 Sep;36(5):574-86. doi: 10.1177/0148607111427040. Epub 2012 Jan 23. PMID 22269899